CLINICAL TRIAL: NCT01624844
Title: Predictive Value of an Ultrasound Model of Measurement of the Dural Sac Volume on the Sensory Level Obtained by Spinal Anesthesia
Brief Title: Predictive Value of Ultrasound Measurement of the Dural Sac Volume on the Sensory Level in Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SG 2012-001
Record Dates: First submitted 2012-06-12; First posted 2012-06-21 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Spinal Anesthesia
Keywords: ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calculation of dural sac volume (Experimental)
  Interventions: Other: Geometrical calculation of dural sac volume

INTERVENTIONS:
Other: Geometrical calculation of dural sac volume — Geometrical calculation of the lumbar dural sac volume following multilevel measurements by ultrasound imaging before spinal anesthesia

SUMMARY:
The purpose of this study is to investigate whether the dural sac volume as determined by a geometrical calculation following multilevel measurements of its transverse area and length by ultrasound imaging, correlates with the intrathecal spread of a single dose of hyperbaric bupivacaine in a non-obstetrical population.

DETAILED DESCRIPTION:
Sensory block extent may be difficult to predict in spinal anesthesia. Many factors influencing the intrathecal spread have been identified. Among the most important factors is the lumbosacral cerebrospinal fluid (CSF) volume and the dimensions of the dural sac. One study using magnetic resonance imaging (MRI) reported significant correlations between CSF volume and sensory block levels following spinal anesthesia. However, unlike ultrasound imaging, MRI can be difficult to obtain in the surgical setting. Although ultrasound imaging of the lumbar spine may not directly determine the CSF volume, multilevel measurements of the transverse area and length of the dural sac by ultrasound imaging followed by a geometrical calculation of its volume could help predict the extent of the intrathecal spread.

Methods: Patients scheduled for elective surgery under spinal anesthesia will be considered for this study. Ultrasound imaging will be achieved in a non-sterile manner with the patient in the sitting position. Spinal imaging will be performed using a low frequency probe. Focus and gain will be optimized. The first images will be made to identify the inter-laminar spaces from T11 to S1. At each level, the area of the dural sac will be measured in short axis using an adjustable ruler built-in the ultrasound monitor. The middle of the inter-laminar spaces will be marked on the patient's skin and the length of the dural sac will be defined as the distance between the middle of T11-12 and L5-S1. The total volume will be geometrically calculated. The L3-L4 space will be localized by triangulation and marked on the patient's skin as the optimal puncture site for spinal anesthesia. The optimal puncture angle will also be determined.

After placement of standard non-invasive monitoring, spinal anesthesia will be performed using 27-G Pencan needle. After aspiration of CSF, a solution of hyperbaric bupivacaine and fentanyl will be injected over a period of 15 seconds. The dose of bupivacaine will be determined by the attendant anaesthesiologist. The aspiration of CSF will be repeated at the end of the injection. Subsequently, the patient will be placed in supine position.

The extent of sensory block will be assessed by loss of pinprick sensation (using a #5.88 Von Frey filament) and loss of cold sensation to ice every 10 minutes until the same sensory level is observed in two consecutive assessments for a minimum period of 30 minutes. The extent of the block will be assessed bilaterally from caudal to cranial direction in the mid-clavicular line beginning at L3. The investigators will consider the peak sensory level as the uppermost blocked dermatome.

Total amount of crystalloids administered, incidence of significant hypotension and bradycardia will be recorded. Time to perform ultrasound measurements and time to discharge will also be noted. Resolution of the motor block will be assessed using the Bromage score at 3.5 hour, 4 and 4.5 hour following the injection of bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients aged 18-80 years
* ASA physical status 1-3

Exclusion Criteria:

* Contraindication to regional anesthesia (coagulopathy, sepsis or local infection at the site of injection, pre-existing neuropathy in the area involved)
* Surgery requiring the use of isobaric bupivacaine (0.5%)
* Allergy to local anesthetics (amide group)
* Anatomic abnormality of the spine (scoliosis, kyphosis)
* Previous spinal surgery
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Geometrical calculation of the lumbar dural sac volume following multilevel measurements by ultrasound imaging | Before spinal anesthesia (Day 0)

SECONDARY OUTCOMES:
Peak sensory level | From injection of bupivacaine until 30 minutes after injection (Day 0)
Time spent for ultrasound imaging measurements | Before spinal anesthesia (Day 0)
Duration of motor block | At 3.5, 4 and 4.5 hours following injection of bupivacaine (Day 0)
Incidence of side-effects related to spinal anesthesia | From spinal injection of bupivacaine until discharge from the hospital (Patients will be followed for the duration of hospital stay, an expected average of 3 days)
Length of stay in the recovery room | From arrival to discharge from the recovery room (Patients will be followed for the duration of stay in the recovery room on the day of surgery, an expected average of one hour)
Length of stay in the hospital | From surgery to discharge from the hospital (Patients will be followed for the duration of hospital stay, an expected average of 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Garneau, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada